CLINICAL TRIAL: NCT02530645
Title: Development and Testing of a Smartphone Application to Reduce Substance Use and Sexual Risk Among Homeless Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #7018
Record Dates: First submitted 2015-08-19; First posted 2015-08-21 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Alcohol Use; Marijuana Use; Sexual Behavior
MeSH Terms: conditions — Alcohol Drinking; Marijuana Use; Sexual Behavior | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OnTrack + BMI (Experimental): Brief motivational interview plus the use of a smartphone application to monitor alcohol and marijuana use and sexual risk behaviors.
  Interventions: Behavioral: OnTrack; Behavioral: Brief Motivational Interviewing
- Treatment as Usual (Active Comparator): Treatment as usual involves substance use/HIV referral and treatment as regularly offered to all participants who report substance use and sexual risk behaviors at Covenant House New York.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: OnTrack
  Arms: OnTrack + BMI
Behavioral: Treatment as Usual
  Arms: Treatment as Usual
Behavioral: Brief Motivational Interviewing
  Arms: OnTrack + BMI

SUMMARY:
A pilot trial (N=60) will be conducted to test the feasibility and preliminary effectiveness of OnTrack (a smartphone application to self-monitor substance use and sexual behaviors among homeless young adults) plus a brief motivational intervention (BMI), in comparison to treatment as usual (TAU) at Covenant House New York (CHNY) for those with substance abuse problems and who engage in risky sex. Following referral, screening, and eligibility determination, 60 participants will complete informed consent and be randomly assigned to one of two conditions: 1) TAU or 2) OnTrack + BMI. All participants will be assessed at baseline, 2 weeks, 4 weeks, and 6 weeks after baseline to evaluate alcohol consumption, marijuana use, HIV sexual risk behaviors, and other relevant variables.

DETAILED DESCRIPTION:
Homeless young adults have high rates of substance abuse and HIV infection and, therefore, developing effective, acceptable, and sustainable interventions to reduce their substance abuse and sexual risk behaviors is of high public health significance.

HealthCall for Smartphone (HealthCall-S) is a smartphone application originally designed for self-monitoring of alcohol use and other HIV-related health behaviors, and receiving personalized feedback on these behaviors among urban substance-abusing HIV primary care patients. Building upon prior HealthCall-S studies, individual qualitative interviews were conducted with 10 homeless young adults (age 18-21 years) at Covenant House New York (CHNY), the largest provider of crisis shelter and services for homeless young adults (age 18-21 years) in NYC. The purpose of the individual interviews was to obtain reactions to various aspects of HealthCall-S and determine how it could be adapted to better suit the needs and interests of homeless young adults. HealthCall-S has since been adapted to target alcohol use, marijuana use, and sexual risk behaviors among homeless young adults and renamed 'OnTrack.' A pilot trial (N=60) will be conducted to test the feasibility and preliminary effectiveness of OnTrack plus a brief motivational intervention (BMI), in comparison to treatment as usual (TAU) at CHNY for those with substance abuse problems and who engage in risky sex. Following referral, screening, and eligibility determination, 60 participants will complete informed consent and be randomly assigned to one of two conditions: 1) TAU or 2) OnTrack + BMI. All participants will be assessed at baseline, 2 weeks, 4 weeks, and 6 weeks after baseline to evaluate alcohol consumption, marijuana use, HIV sexual risk behaviors, and other relevant variables.

ELIGIBILITY:
Inclusion Criteria:

* 18-21 years of age
* Engaged in unprotected vaginal, anal, or oral sex in the past year
* Drank alcohol in the past year
* Used marijuana on 4 or more days in past month

Exclusion Criteria:

* Actively psychotic, suicidal, or homicidal
* Does not speak English
* Has a vision/hearing impairment that would preclude participation
* Has definite plans to leave the greater New York metropolitan area within the study period

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Alcohol use in the last 2 weeks, assessed at baseline and repeatedly so that change can be analyzed | Baseline, 2, 4 (end of treatment), 6 weeks
  As measured by number of drinks per drinking day and percentage of days abstinent.
Marijuana use in the last 2 weeks, assessed at baseline and repeatedly so that change can be analyzed | Baseline, 2, 4 (end of treatment), 6 weeks
  As measured by times used marijuana per day.
HIV sexual risk behavior in the last 2 weeks, assessed at baseline and repeatedly so that change can be analyzed | Baseline, 2, 4 (end of treatment), 6 weeks
  As measured by the number of days the respondent engaged in unprotected sex.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Thompson, Ph.D., Principal Investigator — Columbia University
Locations (1):
- Covenant House New York, New York, New York, United States